CLINICAL TRIAL: NCT00599599
Title: Pilot Intervention for PTSD, Nonadherence, and HIV Risk
Brief Title: Stress-Reducing Interventions in HIV+ Patients: Pilot
Acronym: PEACH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kent State University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Summa Health System (Other)
Responsible Party: Douglas L. Delahanty, Professor, Kent State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R34MH071201-01A1 (NIH); NIMH, 1 R34 MH071201-01A1
Record Dates: First submitted 2008-01-11; First posted 2008-01-24 (Estimated); Last update posted 2009-03-05 (Estimated); Status verified 2009-03

CONDITIONS: Stress Disorders, Post-Traumatic; HIV Infections
Keywords: Prolonged Exposure Therapy; Adherence to HIV Medications; Complementary Therapies
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; HIV Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Prolonged Exposure Therapy.
  Interventions: Behavioral: Prolonged Exposure Therapy
- 2 (No Intervention): Weekly monitoring/Waitlist Control Group.

INTERVENTIONS:
Behavioral: Prolonged Exposure Therapy — Participants will meet with a therapist twice a week for 5 weeks to complete the therapy. If the therapist and participant feel more sessions are needed, an additional 8 sessions will be provided.
  Arms: 1

SUMMARY:
The primary aim of this project is to examine the efficacy of prolonged exposure (PE) therapy at reducing HIV-related PTSD symptoms, increasing adherence to antiretroviral medication regimens, and increasing health-related quality of life (QOL) in HIV+ patients.

DETAILED DESCRIPTION:
HIV+ patients will be randomized to receive either PE therapy (up to 18 possible sessions) or weekly symptom monitoring (described below) and will complete measures of PTSD, adherence, and QOL pre- and post-intervention and at 3- and 6-month follow-up assessments. Secondary analyses will examine the impact of the intervention on disorders commonly comorbid with PTSD (i.e., anxiety, mood, and substance abuse/dependence disorders).

ELIGIBILITY:
Inclusion Criteria:

* Must be HIV+
* Must meet PTSD diagnostic criteria
* Must be taking HIV medications
* Must be able to read and write in English

Exclusion Criteria:

* Current or previous diagnosis of schizophrenia, any current diagnosis with psychotic features, or current suicidal ideation
* Being in a current abusive relationship or ongoing intimate relationship with one's assailant
* Mental retardation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2005-04; Primary Completion 2009-02 (Estimated); Study Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
PTSD symptoms | pre- & post-intervention, 3-month post, & 6-month post

SECONDARY OUTCOMES:
Adherence to HIV medications | pre- & post-intervention, 3-month post, & 6-month post
Health-related Quality of Life | pre- & post-intervention, 3-month post, & 6-month post

CONTACTS AND LOCATIONS:
Overall Officials: Douglas L Delahanty, PhD, Principal Investigator — Kent State University
Locations (2):
- United States (2):
  - Violet's Cupboard, Akron, Ohio
  - AIDS Taskforce of Greater Cleveland, Cleveland, Ohio